CLINICAL TRIAL: NCT03739112
Title: A Randomized, Observer-blind, Active Comparator-controlled, Multicenter, Phase 3 Study to Assess the Efficacy, Safety, and Immunogenicity of a Plant-derived Quadrivalent VLP Influenza Vaccine in Adults 65 Years of Age and Older
Brief Title: Efficacy of a Plant-derived Quadrivalent Virus-like Particle (VLP) Vaccine in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medicago (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-PRO-QVLP-014
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: vaccine; safety; efficacy; plant-made; virus-like particle; hemagglutinin
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Respiratory Tract Diseases; Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: This is a randomized, observer-blind, active comparator-controlled, multicenter, Phase 3 efficacy study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Surveillance personnel is blinded from investigational product injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Quadrivalent VLP Vaccine (Experimental): Participants received one intramuscular (IM) injection of 0.5 mL of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine on Day 0.
  Interventions: Biological: Quadrivalent VLP Vaccine
- Fluarix Quadrivalent® Comparator Vaccine (Active Comparator): Participants received one IM injection of 0.5 mL of 15 μg/strain of the Fluarix Quadrivalent® comparator vaccine on Day 0.
  Interventions: Biological: Fluarix Quadrivalent® Comparator Vaccine

INTERVENTIONS:
Biological: Quadrivalent VLP Vaccine — Single dose of a 30 µg/strain of Quadrivalent VLP Vaccine
  Arms: Quadrivalent VLP Vaccine
Biological: Fluarix Quadrivalent® Comparator Vaccine — Single dose of a 15 μg/strain of Fluarix Quadrivalent® Comparator Vaccine
  Arms: Fluarix Quadrivalent® Comparator Vaccine

SUMMARY:
This Phase 3 study was intended to assess the relative efficacy of the Quadrivalent VLP Influenza Vaccine during the 2018-2019 influenza season compared to a licensed vaccine in elderly adults 65 years of age and older. One dose of VLP Influenza Vaccine (30 μg/strain) or of Comparator (15 μg/strain) was to be administered to 12,738 participants.

DETAILED DESCRIPTION:
This randomized, observer-blind, active-controlled multicenter, Phase 3 study was conducted at multiple sites. The composition of the Quadrivalent VLP Influenza Vaccine used in this study included a mix of recombinant H1, H3, and two B hemagglutinin proteins expressed as VLPs for the 2018-2019 influenza virus strains.

A total of 12,794 healthy male and female participants aged 65 years and older were randomized in a 1:1 ratio into one of two parallel treatment groups, such that 6,396 participants were randomized to receive the Quadrivalent VLP Influenza Vaccine at a dose of 30 μg/strain and 6,398 participants were randomized to receive the comparator. Within the two treatment groups, participants were stratified by site and two age groups (65-74 years of age and 75 years of age and older in a 2:1 ratio).

Participants participated in this study for approximately nine months, during which a first visit was scheduled on Day 0 for screening and vaccine administration.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have read, understood, and signed the informed consent form (ICF) prior to participating in the study; participants must also complete study-related procedures and communicate with the study staff at visits and by phone during the study;
2. Participants must have a body mass index (BMI) ≤35 kg/m^2;
3. Participants are considered by the Investigator to be reliable and likely to cooperate with the assessment procedures and be available for the duration of the study;
4. Male and female participants must be 65 years of age and older at the Screening/Vaccination visit (Visit 1);
5. Participants must be non-institutionalized (e.g. not living in rehabilitation centres or old-age homes; living in an elderly community is acceptable) and have no acute or evolving medical problems prior to study participation and no clinically relevant abnormalities that could jeopardize participant safety or interfere with study assessments, as assessed by the Principal Investigator or sub-Investigator (thereafter referred as Investigator) and determined by medical history, physical examination, and vital signs;

Note: Participants with a pre-existing chronic disease are allowed to participate if the disease is stable and, according to the Investigator's judgment, the condition is unlikely to confound the results of the study or pose additional risk to the participant by participating in the study. Stable disease is generally defined as no new onset or exacerbation of pre-existing chronic disease three months prior to vaccination. Based on the Investigator's judgment, a participant with more recent stabilization of a disease could also be eligible.

Exclusion Criteria:

1. According to the Investigator's opinion, history of an ongoing acute or evolving medical or neuropsychiatric illness. 'Evolving' was defined as:

   * Requiring a new medical or surgical treatment during the three months prior to study vaccine administration unless the criteria outlined in inclusion criterion no. 5 can be met (i.e. the Investigator can justify inclusion based upon the innocuous nature of medical/surgical events and/or treatments);
   * Requiring any significant change in a chronic medication (i.e. drug, dose, frequency) during the three months prior to study vaccine administration due to uncontrolled symptoms or drug toxicity unless the innocuous nature of the medication change meets the criteria outlined in inclusion criterion no. 5 and is appropriately justified by the Investigator.
2. Any medical or neuropsychiatric condition or any history of excessive alcohol use or drug abuse that would render the participant unable to provide informed consent or unable to provide valid safety observations and reporting, including methadone (methadone as treatment for opioid dependence may be acceptable if the participant has been otherwise opioid-free for at least three years);
3. Any autoimmune disease other than hypothyroidism on stable replacement therapy (including, but not limited to rheumatoid arthritis, systemic lupus erythematosus, Crohn's disease, type 1 diabetes, and inflammatory bowel disease) or any confirmed or suspected immunosuppressive condition or immunodeficiency including known or suspected human immunodeficiency virus (HIV), Hepatitis B or C infection, the presence of lymphoproliferative disease;
4. Any history of status asthmaticus or ongoing serious problems with asthma, hospitalization for asthma control, or recurrent asthma episodes requiring medical attention in the last three years (one or more episodes per year);
5. Administration or planned administration of any non-influenza vaccine within 30 days prior to randomization up to blood sampling on Day 21. Immunization on an emergency basis was evaluated case-by-case by the Investigator;
6. Administration of any adjuvanted or investigational influenza vaccine within one year prior to randomization or planned administration prior to the completion of the study;
7. Administration of any 'standard', non-adjuvanted influenza vaccine (e.g. live attenuated trivalent/quadrivalent inactivated influenza vaccine or split trivalent/quadrivalent inactivated influenza vaccine administered by intranasal, intradermal, or IM route) within six months prior to randomization and up to completion of the study;
8. Use of any investigational or non-registered product within 30 days or five half-lives, whichever is longer, prior to randomization or planned use during the study period. Participants may not participate in any other investigational or marketed drug study while participating in this study until after the study;
9. Treatment with systemic glucocorticoids at a dose exceeding 10 mg of prednisone (or equivalent) per day for more than seven consecutive days or for ten or more days in total, within one month of study vaccine administration; any other cytotoxic or immunosuppressant drug, or any immunoglobulin preparation within three months of vaccination and until the completion of the study. Low doses of nasal or inhaled glucocorticoids are allowed. Topical steroids are permitted;
10. Any significant disorder of coagulation including, but not limited to, treatment with warfarin derivatives or heparin. Persons receiving prophylactic anti-platelet medications (e.g. low-dose aspirin [no more than 100 mg/day]), and without a clinically apparent bleeding tendency are eligible. Participants treated with new generation drugs that do not increase the risk of IM bleeding (e.g. clopidogrel) are also eligible;
11. History of allergy to any of the constituents of the Quadrivalent VLP Influenza Vaccine, any components of the active comparator quadrivalent vaccine, or tobacco;
12. History of anaphylactic allergic reactions to plants or plants components (including fruits and nuts);
13. Use of antihistamines within 48 hours prior to study vaccination;
14. Daily use of large doses of medication for pain control or inflammation (e.g. opioids, nonsteroidal anti-inflammatory drugs [NSAIDs]). Use of a singular regular dose either in the morning or at bedtime would not be exclusionary;
15. Use of prophylactic medications (e.g. acetaminophen/paracetamol, aspirin, naproxen, or ibuprofen) within 24 hours of randomization to prevent or pre-empt symptoms due to vaccination;
16. Planned use of influenza antiviral treatment medication before the collection of nasopharyngeal (NP) swabs (e.g. oseltamivir, zanamivir, rapivab);
17. Have a rash, dermatological condition, tattoos, muscle mass, or any other abnormalities at the injection site that may interfere with injection site reaction rating;
18. Participants who have received a blood transfusion within 90 days prior to study vaccination;
19. Participants with abnormal vital signs (systolic blood pressure [BP] ≥ 150 mmHg and/or diastolic BP ≥ 95 mmHg for individuals taking antihypertensive medication and ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg for individuals not taking antihypertensive medication; heart rate [HR] ≤ 45 beats/min and ≥ 100 beats/min) evaluated by an Investigator to be clinically significant. A participant with abnormal vital signs results may be included in the study based on Investigator's judgment (e.g. a resting HR ≤ 45 in highly trained athletes);
20. Presence of any febrile illness (including an oral temperature [OT] ≥ 38.0 ˚C within 24 hours prior to vaccination;
21. Cancer or treatment for cancer within three years prior to study vaccine administration. Persons with a history of cancer who are disease-free without treatment for three years or more are eligible. However, individuals with conditions such as treated and uncomplicated basal cell carcinoma of the skin or non-treated, non-disseminated local prostate cancer may be eligible;
22. Participants identified as an Investigator or employee of the Investigator or clinical site with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse) of the Investigator or any employee of Medicago (or their family members);
23. Participants with a history of Guillain-Barré Syndrome.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12794 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Medicago
Locations (104):
- United States (50):
  - (Site 225) Coastal Clinical Research, Mobile, Alabama
  - (Site 201) Clinical Research Consortium, Tempe, Arizona
  - (Site 213) Advanced Clinical Research, Banning, California
  - (Site 246) Paradigm Clinical Research / Pharmaseek, Redding, California
  - (Site 212) Benckmark Research, Sacramento, California
  - (Site 244) Paradigm Clinical Research Center Inc, San Diego, California
  - (Site 242) Paradigm Clinical Research Centers Inc, Wheat Ridge, Colorado
  - (Site 239) Alliance for Multispeciality Research, Coral Gables, Florida
  - (Site 222) Research Centers of America, Hollywood, Florida
  - (Site 221) St-Johns Center for Clinical Research, Ponte Vedra, Florida
  - (Site 231) QPS-MRA LLC, South Miami, Florida
  - (Site 251) Meridian Clinical Research, Richmond Hill, Georgia
  - (Site 240) Meridian Clinical Research LLC, Savannah, Georgia
  - (Site 223) Clinical Research Atlanta, Stockbridge, Georgia
  - (Site 249) Advanced Clinical Research, Meridian, Idaho
  - (Site 219) Heartland Research Associates LLC, Augusta, Kansas
  - (Site 234) Heartland Research Associates LLC, Newton, Kansas
  - (Site 215) Heartland Research Associates LLC, Wichita, Kansas
  - (Site 235) Heartland Research Associates LLC, Wichita, Kansas
  - (Site 241) Central Kentucky Reserach Associates, Lexington, Kentucky
  - (Site 203) Benchmark Research, Metairie, Louisiana
  - (Site 227) Sundande Clinical Research, St Louis, Missouri
  - (Site 226) Meridian Clinical Research LLC, Norfolk, Nebraska
  - (Site 211) Meridian Clinical Research, Omaha, Nebraska
  - (Site 209) United Medical Associates, Binghamton, New York
  - (Site 217) Regional Clinical Research inc, Endwell, New York
  - (Site 237) PMG Research of Cary LLC, Cary, North Carolina
  - (Site 230) PMG Research of Charlotte LLC, Charlotte, North Carolina
  - (Site 205) PMG Research of Rocky Mount LLC, Rocky Mount, North Carolina
  - (Site 236) PMG Research, Statesville, North Carolina
  - (Site 228) Research of Winston-Salem, Winston-Salem, North Carolina
  - (Site 233) Sterling Research Group, Cincinnati, Ohio
  - (Site 208) Sterling Research Group, Cincinnati, Ohio
  - (Site 245) Rapid Medical Research, Cleveland, Ohio
  - (Site 202) Aventiv Research Inc, Columbus, Ohio
  - (Site 207) Lynn Institute of Norman, Norman, Oklahoma
  - (Site 238) Tekton Research, Oklahoma City, Oklahoma
  - (Site 216) PMG Research of Charleston LLC, Mt. Pleasant, South Carolina
  - (Site 248) Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - (Site 201) Meridian Clinical Research, Dakota Dunes, South Dakota
  - (Site 247) New orleans Center for Clinical Research, Knoxville, Tennessee
  - (Site 206) Benchmark Research, Austin, Texas
  - (Site 218) Tekton Research Inc, Austin, Texas
  - (Site 214) Ventavia Research Group LLC, Fort Worth, Texas
  - (Site 224) Benchmark Research, Fort Worth, Texas
  - (Site 232) Benchmark Research, San Angelo, Texas
  - (Site 250) Clinical Trials of Texas Inc, San Antonio, Texas
  - (Site 204) Jean Brown Research, Salt Lake City, Utah
  - (Site 220) Advanced Clinical Research, West Jordan, Utah
  - (Site 229) Clinical Research Associates of Tidewater, Norfolk, Virginia
- Canada (13):
  - (Site 106) Colchester Research Group, Truro, Nova Scotia
  - (Site 113) Dawson Road Family Medical Clinic, Guelph, Ontario
  - (Site 110) Manna Research Inc., Toronto, Ontario
  - (Site 103) Q & T Recherche Chicoutimi, Chicoutimi, Quebec
  - (Site 105) Q & T Outaouais, Gatineau, Quebec
  - (Site 107) Manna Research Inc., Lévis, Quebec
  - (Site 109) Manna Research Inc. (Mirabel), Mirabel, Quebec
  - (Site 108) Manna Research, Pointe-Claire, Quebec
  - (Site 102) CHU de Québec - Université Laval, Québec, Quebec
  - (site 101) Centre de Recherche St-Louis, Québec, Quebec
  - (Site 110) Alpha Recherche Clinique, Québec, Quebec
  - (Site 104) Q & T Recherche Sherbrooke, Sherbrooke, Quebec
  - (Site 112) Medexa Recherche, Victoriaville, Quebec
- Finland (10):
  - (Site 309) Espoo Vaccine Research Clinic, Espoo
  - (Site 303) Helsinki South Vaccine Research Clinic, Helsinki
  - (Site 308) Helsinki East Vaccine Research Center, Helsinki
  - (Site 301) Jarvenpaa Vaccine Research Clinic, Jarvenpaa
  - (Site 306) Kokkola Vaccine Research Clinic, Kokkola
  - (Site 304) Oulu Vaccine Research Clinic, Oulu
  - (Site 302) Tampere University Vaccine Research Center, Pori
  - (Site 305) Seinaejoki Vaccine Research Clinic, Seinäjoki
  - (Site 310) Tampere Vaccine Research Clinic, Tampere
  - (Site 307) Turku Vaccine Research Center, Turku
- Germany (24):
  - (Site 410) Emovis GmbH, Berlin
  - (Site 418) Klinische Forschung Berlin GbR, Berlin
  - (Site 422) Synexus Clinical Research GmbH, Berlin
  - (Site 402) Synexus Clinical research GmbH, Bochum
  - (Site 409) Gemeinschaftspraxis Dr. med Kleinecke-Pohl, Cologne
  - (Site 401) Cardiologicum Dresden & Pirna, Dresden
  - (Site 406) Diabetologische Germeinschafts praxis Faulman, Dresden
  - (Site 405) Doktor Markus Faghih, Essen
  - (Site 407) Klinisches Forschungszentrum Dr. Hagemann am Hausarztzer, Essen
  - (Site 417) Medizentrum Essen-Borbeck, Essen
  - (Site 414) Unterfrintroper Hausarztzentrum Klinische Forschung, Essen
  - (SIte 404) Synexus Clinical Reserach GmbH, Frankfurt
  - (Site 411) MedicoKIT GmbH, Goch
  - (Site 425) Clinical Research Hamburg, Hamburg
  - (Site 403) Praxis Dr. Med Cornelia Brauer, Hamburg
  - (Site 408) Germeinsschaftspraxis Dr. med Christiane Klein/Minnich, Künzing
  - (Site 421) SIBAmed Studienzentrum GmbH, Leipzig
  - (Site 420) Synexus Clinical Research GmbH, Leipzig
  - (Site 423) centrum fuer Diagnostik und Gesundheit, Munich
  - (Site 413) Dr. Ingomar F.K. Naudts MD Office, Rodgau
  - (Site 415) Praxisgemeinschaft Stuhr-Brinkum, Stuhr
  - (Site 416) Praxis Dr. med Joachim Sauter, Wangen
  - (Site 412) MALU-Medizinische Studien GmbH, Wardenburg
  - (Site 424) Medislim GmbH, Weinheim
- Thailand (7):
  - (Site 603) Ramathibodi Hospital, Mahid - Division of Infectious Disease, Bangkok
  - (Site 606) Faculty of Tropical Medicine, Mahidol University, Bangkok
  - (Site 608) Phramongkutklao Hospital, Bangkok
  - (Site 609) Division of Tropical Pediatrics, Bangkok
  - (Site 601) Faculty of Medicine, Chiang Mai University, Chiang Mai
  - (Site 607) Srinagarind Hospital Khon Kaen University, Khon Kaen
  - (Site 605) Golden Jubilee Medical Center, Nakhon Pathom

REFERENCES:
- [Result] Ward BJ, Makarkov A, Seguin A, Pillet S, Trepanier S, Dhaliwall J, Libman MD, Vesikari T, Landry N. Efficacy, immunogenicity, and safety of a plant-derived, quadrivalent, virus-like particle influenza vaccine in adults (18-64 years) and older adults (>/=65 years): two multicentre, randomised phase 3 trials. Lancet. 2020 Nov 7;396(10261):1491-1503. doi: 10.1016/S0140-6736(20)32014-6. Epub 2020 Oct 13. PMID 33065035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized in a 1:1 ratio to receive the Quadrivalent virus-like particle (VLP) Influenza Vaccine at a dose of 30 μg/strain or the active comparator.
Pre-assignment Details: Participants aged 65 years or older with no acute or evolving medical problems were assessed.
Groups:
- Quadrivalent (30 μg) VLP Vaccine: Participants received one intramuscular (IM) injection of 0.5 mL of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine on Day 0.
- Active Comparator (Fluarix): Participants received one IM injection of 0.5 mL of 15 μg/strain of the Fluarix Quadrivalent® comparator vaccine on Day 0.
Period: Overall Study
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Started | 6396 | 6398
Vaccinated | 6365 | 6373
Completed | 6196 | 6222
Not Completed | 200 | 176
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 38 | 19
Not completed — Lost to Follow-up | 31 | 33
Not completed — Protocol Deviation | 12 | 9
Not completed — Physician Decision | 1 | 0
Not completed — Death (Classified as Withdrawn from the Study by the Investigator as a Result of Death) | 12 | 16
Not completed — Site went on hold | 65 | 67
Not completed — Other than specified | 8 | 5
Not completed — Randomized but not vaccinated | 31 | 25

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) was defined as all participants who received either the Quadrivalent VLP Influenza Vaccine or the active comparator. Participants that were non-compliant to protocol/Good Clinical Practice (GCP), as per investigator, were excluded from analysis.
Groups:
- Quadrivalent (30 μg) VLP Vaccine: Participants received one IM injection of 0.5 mL of 30 μg/strain of the Quadrivalent VLP Influenza Vaccine on Day 0.
- Total: Total of all reporting groups
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix) | Total
Number analyzed (Participants) | 6352 | 6366 | 12718
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (5.67) | 72.2 (5.70) | 72.2 (5.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3552 | 3561 | 7113
  Male | 2800 | 2805 | 5605
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 202 | 195 | 397
  Not Hispanic or Latino | 6135 | 6161 | 12296
  Unknown or Not Reported | 15 | 10 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19 | 13 | 32
  Asian | 305 | 299 | 604
  Native Hawaiian or Other Pacific Islander | 5 | 5 | 10
  Black or African American | 248 | 265 | 513
  White | 5767 | 5773 | 11540
  More than one race | 6 | 10 | 16
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Occurrences of Protocol-Defined Influenza-Like Illness (ILI) Due to Any Laboratory-Confirmed Influenza Strains
Description: Occurrences of laboratory-confirmed ILI caused by any influenza viral strains was measured by reverse transcriptase polymerase chain reaction (RT-PCR). A participant was considered to have protocol-defined ILI if the participant met at least one of the following pre-defined respiratory symptoms: sore throat, cough, sputum production, wheezing, or difficulty breathing and at least one of the following systemic symptoms: fever (defined as a temperature > 37.2 °C or > 99.0 °F), chills, tiredness, headache or myalgia. The number of laboratory-confirmed ILI cases caused by any influenza strains are reported.
Time Frame: Day 14 (post-vaccination) up to ~9 months
Population: The Per protocol (PP) set consisted of the participants who participated in the study until at least the end of the peak period or for at least five months or until the end of the surveillance period.
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 5996 | 6026
Number of cases | 118 | 130
Statistical Analysis 1: Comparison: Quadrivalent (30 μg) VLP Vaccine vs Active Comparator (Fluarix); Test type: Non-Inferiority — Non-inferiority was concluded if the lower limit of the two-sided 95% confidence interval (CI) for relative vaccine efficacy (VE) was > -20%; percent VE = 8.8, 95% CI 2-sided [-16.7 to 28.7] — VE of VLP vaccine versus Fluarix = (1-ARVv/ARVc) x 100% where ARVv = attack rate in participants vaccinated with the Quadrivalent VLP Influenza vaccine and ARVc = attack rate in participants vaccinated with an active Fluarix

2. Secondary Outcome: Number of Occurrences of Laboratory Confirmed Protocol-Defined Influenza-Like Illness (ILI) Caused by Vaccine-Matched Influenza Strains
Description: Occurrences of protocol-defined ILI due to laboratory-confirmed influenza caused by influenza viral types/subtypes that were matched (and/or antigenically similar) to the strains covered in the vaccine formulation was measured by sequential RT-PCR & serotyping. The vaccine-matched strains included: homologous A/Michigan/45/2015 [H1N1], homologous A/Singapore/INFIMH-16-0019/2016 [H3N2], homologous B/Colorado/06/2017 and homologous B/Phuket/3073/2013) covered in the vaccine formulation. A participant was considered to have protocol-defined ILI if the participant met at least one of the following pre-defined respiratory symptoms: sore throat, cough, sputum production, wheezing, or difficulty breathing and at least one of the following systemic symptoms: fever (defined as a temperature > 37.2 °C or > 99.0 °F), chills, tiredness, headache or myalgia. The number of laboratory-confirmed ILI cases caused by vaccine-matched influenza strains (all matched strains) are reported.
Time Frame: Day 14 (post-vaccination) up to ~9 months
Population: PP set.
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 5996 | 6026
Number of cases | 42 | 46

3. Secondary Outcome: Number of Occurrences of Protocol-Defined Respiratory Illness Due to Any Laboratory-Confirmed Influenza Strains
Description: Occurrences of protocol-defined respiratory illness due to laboratory-confirmed influenza strain (matched, mismatched, and un-typed) was measured by sequential RT-PCR. A protocol-defined respiratory illness was determined by the occurrence of at least 1 of the following respiratory symptoms: sneezing, stuffy nose, sore throat, cough, sputum production, wheezing, or difficulty breathing. The number of protocol-defined respiratory illness cases caused by any laboratory-confirmed influenza strain (matched, mismatched, and un-typed) are reported.
Time Frame: Day 14 (post-vaccination) up to ~9 months
Population: PP set.
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 5996 | 6026
Number of cases | 148 | 167

4. Secondary Outcome: Number of Occurrences of Protocol-Defined Respiratory Illness Vaccine Caused by Vaccine-Matched Influenza Strains
Description: Occurrences of protocol-defined respiratory illness vaccine caused by vaccine-matched influenza strains was measured by sequential RT-PCR & serotyping. The vaccine-matched strains included: homologous A/Michigan/45/2015 [H1N1], homologous A/Singapore/INFIMH-16-0019/2016 [H3N2], homologous B/Colorado/06/2017 and homologous B/Phuket/3073/2013. The protocol-defined respiratory illness was determined by the occurrence of at least 1 of the following respiratory symptoms: sneezing, stuffy nose, sore throat, cough, sputum production, wheezing, or difficulty breathing. The number of protocol-defined respiratory illness cases caused by one or more vaccine-matched strains are reported.
Time Frame: Day 14 (post-vaccination) up to ~9 months
Population: PP set.
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 5996 | 6026
Number of cases | 50 | 55

5. Secondary Outcome: Number of Occurrences of Protocol-Defined ILI
Description: Occurrences of protocol-defined ILI that were confirmed or not by laboratory testing were assessed. A participant was considered to have protocol-defined ILI if the participant met at least one of the following pre-defined respiratory symptoms: sore throat, cough, sputum production, wheezing, or difficulty breathing and at least one of the following systemic symptoms: fever (defined as a temperature > 37.2 °C or > 99.0 °F), chills, tiredness, headache or myalgia. The number of protocol-defined ILI cases (confirmed or not) are reported.
Time Frame: Day 14 (post-vaccination) up to ~9 months
Population: PP set.
Measure: Number; unit: Number of cases
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 5996 | 6026
Number of cases | 1249 | 1243

6. Secondary Outcome: Number of Participants With at Least One Immediate Complaints
Description: Immediate complaints were defined as any solicited local or systemic reactions. Solicited local reactions included: erythema, swelling, and pain at the injection site) and solicited systemic reactions included: fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck.
Time Frame: 15 minutes post vaccination
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 272 | 184

7. Secondary Outcome: Number of Participants With at Least One Solicited Local and Systemic Reactions
Description: Participants were monitored for both solicited local reactions (erythema, swelling, and pain at the injection site) and solicited systemic reactions (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck) from the time of vaccination through Day 7. Any solicited local or systemic immediate complaint was also included.
Time Frame: Day 0 (post-vaccination) to Day 7
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants
  Solicited Local Reactions | 1954 | 1460
  Solicited Systemic Reactions | 1682 | 1497

8. Secondary Outcome: Number of Participants With ≥ Severe Solicited Local and Systemic Reaction
Description: Participants were monitored for both solicited local reactions (erythema, swelling, and pain at the injection site) and solicited systemic reactions (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in the axilla, and swelling in the neck). The intensity of the solicited reactions was graded as mild (1)-easily tolerated and does not interfere with usual activity; moderate (2)-interferes with daily activity, but the participant is still able to function; severe (3)-incapacitating and the participant is unable to work or complete usual activity or potentially life threatening; (4)-likely to be life-threatening if not treated in a timely manner, according to the Food and Drug Administration (FDA) Guidance for Industry. ≥ Severe events included severe and potentially life-threatening events. Any ≥severe solicited reactions are reported.
Time Frame: Day 0 (post-vaccination) to Day 7
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 47 | 62

9. Secondary Outcome: Number of Participants With ≥ Severe Related Solicited Reactions
Description: Participants were monitored for both solicited local reactions (erythema, swelling, & pain at the injection site) & solicited systemic reactions (fever, headache, fatigue, muscle aches, joint aches, chills, a feeling of general discomfort, swelling in axilla, & swelling in neck). The intensity of solicited reactions was graded as mild (1)-easily tolerated and does not interfere with usual activity; moderate (2)-interferes with daily activity, but the participant is still able to function; severe (3)-incapacitating and the participant is unable to work or complete usual activity or potentially life threatening; (4)-likely to be life-threatening if not treated in a timely manner, according to the FDA Guidance for Industry. ≥ Severe events included severe and potentially life-threatening events. Any ≥severe related (possibly related, probably related, and definitely related to the study treatments [as defined by investigator]) solicited events are reported.
Time Frame: Day 0 (post-vaccination) to Day 7
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 28 | 51

10. Secondary Outcome: Number of Participants With Unsolicited Treatment-Emergent Adverse Events (TEAEs)
Description: Participants were monitored for unsolicited TEAEs (e.g., nasopharyngitis, upper respiratory tract infection, headache, and pain). An adverse event (AE) or adverse experience was defined as any untoward medical occurrence in a participant or clinical investigation participant who received study drug, with or without a causal relationship with the treatment. An AE was considered treatment-emergent if it began on or after the date and time of Study Day 0 vaccination.
Time Frame: Day 0 (post-vaccination) to Day 21
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 849 | 824

11. Secondary Outcome: Number of Participants With ≥ Severe Unsolicited TEAEs
Description: Participants were monitored for unsolicited TEAEs (e.g., nasopharyngitis, upper respiratory tract infection, headache, and pain). AE: any untoward medical occurrence in a participant or clinical investigation participant who received study drug, with or without a causal relationship with the treatment. An AE was considered treatment-emergent if it began on or after the date and time of Study Day 0 vaccination. The intensity of the solicited reactions was graded as mild (1)-easily tolerated and does not interfere with usual activity; moderate (2)-interferes with daily activity, but the participant is still able to function; severe (3)-incapacitating and the participant is unable to work or complete usual activity or potentially life threatening; (4)-likely to be life-threatening if not treated in a timely manner, according to the FDA Guidance for Industry. ≥ severe events included severe and potentially life-threatening events. Any ≥ severe unsolicited reactions are reported.
Time Frame: Day 0 (post-vaccination) to Day 21
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 33 | 34

12. Secondary Outcome: Number of Participants With ≥ Severe Related Unsolicited Reactions
Description: Participants were monitored for unsolicited TEAEs (e.g., nasopharyngitis, upper respiratory tract infection, headache, & pain). AE: any untoward medical occurrence in a participant who received study drug, with or without a causal relationship with treatment. An AE was considered treatment-emergent if it began on or after date & time of Study Day 0 vaccination. Intensity of solicited reactions was graded as mild (1) easily tolerated & not interfere with usual activity; moderate (2) interferes with daily activity, but participant still able to function; severe (3) incapacitating & participant unable to work/complete usual activity/ potentially life threatening; (4) likely to be life-threatening if not treated in a timely manner, according to FDA Guidance for Industry. ≥ severe events included severe & potentially life-threatening events. Any ≥severe related (possibly, probably, & definitely related to study treatments [as defined by investigator]) unsolicited events are reported.
Time Frame: Day 0 (post-vaccination) to Day 21
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 1 | 3

13. Secondary Outcome: Number of Participants With at Least One Serious Adverse Event (SAE)
Description: An AE was any untoward medical occurrence in a participant who received study drug, with or without a causal relationship with treatment. An SAE was an AE that resulted in death, was life threatening, resulted in a persistent or significant disability or incapacity, resulted in or prolonged an existing hospitalization, was a congenital anomaly or birth defect, or was another important medical event.
Time Frame: Day 0 to ~9 months
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 263 | 266

14. Secondary Outcome: Number of Occurrences of Death
Description: The number of participants who died during the study was assessed.
Time Frame: Day 0 up to ~9 months
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 12 | 17

15. Secondary Outcome: Number of Participants Who Withdrew Due to an AE
Description: An AE or adverse experience was defined as any untoward medical occurrence in a participant or clinical investigation participant who received study drug, with or without a causal relationship with the treatment. An AE can be any favorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to a medicinal product.
Time Frame: Day 0 up to ~9 months
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 15 | 20

16. Secondary Outcome: Number of Participants With at Least One New Onset Chronic Diseases (NOCDs)
Description: All NOCDs that may plausibly have an allergic, autoimmune or inflammatory component were reported. Plausibility should be interpreted broadly however; the only clear exceptions were degenerative conditions such as osteoarthritis, age-related physiologic changes and life-style diseases. In this context, most cancers, cardiac conditions and kidney diseases should be reported. NOCDs were collected from vaccination on Day 0 to the end of the surveillance period.
Time Frame: Day 0 up to ~9 months
Population: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 6352 | 6366
Participants | 36 | 23

17. Secondary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HI) Antibody Response for Each Homologous and Heterologous Influenza Strain
Description: GMTs were measured using a HI assay for the homologous strains: H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013, and the heterologous strains: H1N1 = A/Brisbane/59/2007; H3N2 = A/Uruguay/716/2007; B/Malaysia = B/Malaysia/2506/2004; B/Florida = B/Florida/4/2006.
Time Frame: Baseline (Day 0), Day 21
Population: The Immunogenicity Per Protocol (IPP) set consisted of a subset of participants who participated in the immunogenicity portion of the study and who had a Day 21 immunogenicity sample collection.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
Titers
  Homologous Strain (H1N1): Day 0 | 43.8 [36.3 to 52.7] | 36.3 [30.0 to 43.9]
  Homologous Strain (H1N1): Day 21 | 88.9 [73.7 to 107.2] | 146.8 [121.4 to 177.7]
  Homologous Strain (H3N2): Day 0 | 31.1 [25.5 to 37.8] | 30.9 [25.3 to 37.8]
  Homologous Strain (H3N2): Day 21 | 79.5 [65.2 to 97.1] | 90.2 [73.7 to 110.5]
  Homologous Strain (B/Colorado): Day 0 | 15.5 [13.3 to 18.1] | 13.2 [11.3 to 15.5]
  Homologous Strain (B/Colorado): Day 21 | 23.0 [19.3 to 27.4] | 51.7 [43.3 to 61.8]
  Homologous Strain (B/Phuket): Day 0 | 24.4 [20.8 to 28.7] | 22.6 [19.2 to 26.6]
  Homologous Strain (B/Phuket): Day 21 | 45.0 [37.8 to 53.5] | 75.5 [63.3 to 90.1]
  Heterologous Strain (H1N1): Day 0 | 15.5 [13.6 to 17.6] | 13.5 [11.8 to 15.4]
  Heterologous Strain (H1N1): Day 21 | 16.6 [14.3 to 19.2] | 32.4 [28.0 to 37.6]
  Heterologous Strain (H3N2): Day 0 | 19.5 [16.4 to 23.3] | 22.6 [18.9 to 27.1]
  Heterologous Strain (H3N2): Day 21 | 32.4 [27.1 to 38.6] | 46.6 [38.9 to 55.8]
  Heterologous Strain (B/Malaysia): Day 0 | 12.6 [11.0 to 14.5] | 11.4 [10.0 to 13.1]
  Heterologous Strain (B/Malaysia): Day 21 | 15.9 [13.6 to 18.7] | 34.8 [29.5 to 41.0]
  Heterologous Strain (B/Florida): Day 0 | 22.5 [19.2 to 26.4] | 20.6 [17.5 to 24.2]
  Heterologous Strain (B/Florida): Day 21 | 38.0 [32.2 to 44.8] | 72.1 [61.0 to 85.2]

18. Secondary Outcome: Percentage of Participants With Seroconversion Measured by HI Antibody Response for Each Homologous and Heterologous Strain
Description: The percentage of participants in a given treatment group with either a ≥ 4-fold increase in reciprocal HI titers between Day 0 and Day 21 or a rise of undetectable HI titer (i.e. < 10) pre-vaccination (Day 0) to an HI titer of ≥ 40 on Day 21 was measured using an HI assay for the homologous strains: H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013, and the heterologous strains: H1N1 = A/Brisbane/59/2007; H3N2 = A/Uruguay/716/2007; B/Malaysia = B/Malaysia/2506/2004; B/Florida = B/Florida/4/2006.
Time Frame: Day 0 (pre-vaccination) to Day 21
Population: IPP set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
percentage of participants
  Homologous Strain (H1N1) | 15.5 [10.9 to 21.2] | 40.7 [33.8 to 47.9]
  Homologous Strain (H3N2) | 25.2 [19.5 to 31.7] | 28.1 [22.0 to 34.9]
  Homologous Strain (B/Colorado) | 10.2 [6.4 to 15.2] | 38.2 [31.4 to 45.3]
  Homologous Strain (B/Phuket) | 16.5 [11.7 to 22.3] | 34.7 [28.1 to 41.7]
  Heterologous Strain (H1N1) | 0.5 [0.0 to 2.7] | 24.1 [18.4 to 30.7]
  Heterologous Strain (H3N2) | 10.7 [6.8 to 15.7] | 14.6 [10.0 to 20.3]
  Heterologous Strain (B/Malaysia) | 5.3 [2.7 to 9.4] | 30.7 [24.3 to 37.6]
  Heterologous Strain (B/Florida) | 12.1 [8.0 to 17.4] | 37.7 [30.9 to 44.8]

19. Secondary Outcome: Percentage of Participants With Seroprotection Measured by HI Antibody Response for Each Homologous and Heterologous Strain
Description: The percentage of participants in a given treatment group attaining a reciprocal HI titer of ≥ 40 on Day 21 (the percentage of vaccine recipients with a serum HI titer of at least 1:40 following vaccination) was measured using an HI assay for homologous strains: H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013, and the heterologous strains: H1N1 = A/Brisbane/59/2007; H3N2 = A/Uruguay/716/2007; B/Malaysia = B/Malaysia/2506/2004; B/Florida = B/Florida/4/2006.
Time Frame: Baseline (Day 0), Day 21
Population: IPP set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
percentage of participants
  Homologous Strain (H1N1): Day 0 | 57.3 [50.2 to 64.1] | 52.8 [45.6 to 59.9]
  Homologous Strain (H1N1): Day 21 | 77.2 [70.8 to 82.7] | 87.9 [82.6 to 92.1]
  Homologous Strain (H3N2): Day 0 | 48.5 [41.5 to 55.6] | 52.8 [45.6 to 59.9]
  Homologous Strain (H3N2): Day 21 | 72.3 [65.7 to 78.3] | 78.4 [72.0 to 83.9]
  Homologous Strain (B/Colorado): Day 0 | 28.6 [22.6 to 35.3] | 22.1 [16.5 to 28.5]
  Homologous Strain (B/Colorado): Day 21 | 40.3 [33.5 to 47.3] | 62.3 [55.2 to 69.1]
  Homologous Strain (B/Phuket): Day 0 | 46.6 [39.6 to 53.7] | 38.7 [31.9 to 45.8]
  Homologous Strain (B/Phuket): Day 21 | 64.1 [57.1 to 70.6] | 79.4 [73.1 to 84.8]
  Heterologous Strain (H1N1): Day 0 | 21.8 [16.4 to 28.1] | 18.1 [13.0 to 24.2]
  Heterologous Strain (H1N1): Day 21 | 22.8 [17.3 to 29.2] | 49.2 [42.1 to 56.4]
  Heterologous Strain (H3N2): Day 0 | 35.4 [28.9 to 42.4] | 40.2 [33.3 to 47.4]
  Heterologous Strain (H3N2): Day 21 | 50.0 [43.0 to 57.0] | 63.8 [56.7 to 70.5]
  Heterologous Strain (B/Malaysia): Day 0 | 22.8 [17.3 to 29.2] | 17.6 [12.6 to 23.6]
  Heterologous Strain (B/Malaysia): Day 21 | 30.1 [23.9 to 36.9] | 53.8 [46.6 to 60.8]
  Heterologous Strain (B/Florida): Day 0 | 37.4 [30.8 to 44.4] | 31.2 [24.8 to 38.1]
  Heterologous Strain (B/Florida): Day 21 | 58.7 [51.7 to 65.5] | 76.9 [70.4 to 82.6]

20. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of HI Antibody Response for Each Homologous and Heterologous Strain
Description: GMFR, the geometric mean of the ratio of GMTs (Day 21/Day 0), was measured using an HI assay homologous strains: H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013, and the heterologous strains: H1N1 = A/Brisbane/59/2007; H3N2 = A/Uruguay/716/2007; B/Malaysia = B/Malaysia/2506/2004; B/Florida = B/Florida/4/2006.
Time Frame: Baseline (Day 0), Day 21
Population: IPP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
Ratio
  Homologous Strain (H1N1) | 2.1 [1.8 to 2.4] | 3.9 [3.4 to 4.5]
  Homologous Strain (H3N2) | 2.6 [2.2 to 3.0] | 2.9 [2.5 to 3.4]
  Homologous Strain (B/Colorado) | 1.5 [1.3 to 1.8] | 3.8 [3.3 to 4.4]
  Homologous Strain (B/Phuket) | 1.9 [1.6 to 2.1] | 3.3 [2.9 to 3.8]
  Heterologous Strain (H1N1) | 1.1 [1.0 to 1.2] | 2.4 [2.2 to 2.6]
  Heterologous Strain (H3N2) | 1.6 [1.5 to 1.8] | 2.1 [1.9 to 2.3]
  Heterologous Strain (B/Malaysia) | 1.3 [1.1 to 1.4] | 3.0 [2.7 to 3.4]
  Heterologous Strain (B/Florida) | 1.7 [1.5 to 1.9] | 3.4 [3.0 to 3.9]

21. Secondary Outcome: GMTs of Microneutralization (MN) Antibody Response for Each Homologous Strain
Description: GMTs were measured using an MN assay for homologous strains:H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013.
Time Frame: Baseline (Day 0), Day 21
Population: IPP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
Titers
  H1N1: Day 0 | 501.4 [420.6 to 597.8] | 511.2 [427.5 to 611.3]
  H1N1: Day 21 | 1120.7 [926.3 to 1355.9] | 1807.0 [1488.6 to 2193.6]
  H3N2: Day 0 | 227.4 [194.9 to 265.3] | 240.1 [205.3 to 280.8]
  H3N2: Day 21 | 558.5 [461.2 to 676.3] | 437.0 [359.7 to 531.0]
  B/Colorado: Day 0 | 62.7 [54.1 to 72.6] | 55.1 [47.5 to 64.0]
  B/Colorado: Day 21 | 124.1 [105.4 to 146.2] | 193.1 [163.5 to 228.1]
  B/Phuket: Day 0 | 50.5 [44.4 to 57.6] | 45.8 [40.1 to 52.3]
  B/Phuket: Day 21 | 98.2 [85.7 to 112.6] | 143.4 [124.8 to 164.7]

22. Secondary Outcome: Percentage of Participants With Seroconversion Measured by MN Antibody Response for Each Homologous Strain
Description: The percentage of participants in a given treatment group with either a ≥ 4-fold increase in reciprocal MN titers between Day 0 and Day 21 or a rise of undetectable MN titer (i.e. 7.1) pre-vaccination (Day 0) to an MN titer of ≥ 28.3 at Day 21 post-vaccination were measured using an MN assay for homologous strains: H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013.
Time Frame: Day 0 (pre-vaccination) to Day 21
Population: IPP set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
percentage of participants
  H1N1 | 25.7 [19.9 to 32.3] | 43.2 [36.2 to 50.4]
  H3N2 | 36.4 [29.8 to 43.4] | 26.6 [20.6 to 33.3]
  B/Colorado | 19.9 [14.7 to 26.0] | 43.7 [36.7 to 50.9]
  B/Phuket | 19.4 [14.2 to 25.5] | 41.2 [34.3 to 48.4]

23. Secondary Outcome: GMFR of MN Antibody Response for Each Homologous Strain
Description: GMFR, the geometric mean of the ratio of GMTs (Day 21/Day 0), was measured using an MN assay for H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013.
Time Frame: Baseline (Day 0), Day 21
Population: IPP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
Ratio
  H1N1 | 2.2 [1.9 to 2.6] | 3.5 [3.0 to 4.1]
  H3N2 | 2.4 [2.1 to 2.8] | 1.8 [1.6 to 2.1]
  B/Colorado | 2.0 [1.8 to 2.3] | 3.4 [3.0 to 3.9]
  B/Phuket | 2.0 [1.8 to 2.2] | 3.1 [2.8 to 3.4]

24. Secondary Outcome: Geometric Mean Areas (GMA) of Single Radial Hemolysis (SRH) Antibody Response for Each Homologous Strain
Description: GMA was measured using an SRH assay for homologous strains: H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013.
Time Frame: Baseline (Day 0), Day 21
Population: IPP set.
Measure: Geometric Mean (95% Confidence Interval); unit: mm^2
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
mm^2
  H1N1: Day 0 | 23.8 [20.4 to 27.7] | 20.7 [17.7 to 24.2]
  H1N1: Day 21 | 38.7 [34.7 to 43.1] | 48.9 [43.8 to 54.6]
  H3N2: Day 0 | 6.3 [5.1 to 7.9] | 5.1 [4.1 to 6.3]
  H3N2: Day 21 | 21.9 [17.2 to 28.0] | 13.2 [10.3 to 17.0]
  B/Colorado: Day 0 | 33.7 [28.1 to 40.3] | 29.2 [24.3 to 35.1]
  B/Colorado: Day 21 | 54.1 [47.3 to 61.8] | 61.0 [53.3 to 69.9]
  B/Phuket: Day 0 | 21.5 [17.7 to 26.0] | 20.4 [16.8 to 24.8]
  B/Phuket: Day 21 | 38.8 [33.5 to 44.9] | 50.2 [43.3 to 58.3]

25. Secondary Outcome: Percentage of Participants With Seroconversion Measured by SRH Antibody Response for Each Homologous Strain
Description: The percentage of participants in a given treatment group showing at least 50 % increase in GMA between Days 0 and 21 were measured using an SRH assay for homologous strains: H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013.
Time Frame: Day 0 (pre-vaccination) to Day 21
Population: IPP set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
percentage of participants
  H1N1 | 34.0 [27.5 to 40.9] | 55.3 [48.1 to 62.3]
  H3N2 | 45.1 [38.2 to 52.2] | 34.7 [28.1 to 41.7]
  B/Colorado | 32.0 [25.7 to 38.9] | 49.7 [42.6 to 56.9]
  B/Phuket | 35.9 [29.4 to 42.9] | 52.3 [45.1 to 59.4]

26. Secondary Outcome: Percentage of Participants With Seroprotection Measured by SRH Antibody Response for Each Homologous Strain
Description: The percentage of participants in a given treatment group attaining an area ≥ 25 mm^2 following vaccination (Day 21) were measured using an SRH assay for homologous strains: H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013.
Time Frame: Baseline (Day 0), Day 21
Population: IPP set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
percentage of participants
  H1N1: Day 0 | 56.8 [49.7 to 63.7] | 51.8 [44.6 to 58.9]
  H1N1: Day 21 | 77.7 [71.4 to 83.2] | 89.4 [84.3 to 93.3]
  H3N2: Day 0 | 27.7 [21.7 to 34.3] | 23.6 [17.9 to 30.1]
  H3N2: Day 21 | 63.6 [56.6 to 70.2] | 51.8 [44.6 to 58.9]
  B/Colorado: Day 0 | 71.8 [65.2 to 77.9] | 69.8 [63.0 to 76.1]
  B/Colorado: Day 21 | 87.9 [82.6 to 92.0] | 89.4 [84.3 to 93.3]
  B/Phuket: Day 0 | 63.6 [56.6 to 70.2] | 60.8 [53.7 to 67.6]
  B/Phuket: Day 21 | 76.2 [69.8 to 81.9] | 87.9 [82.6 to 92.1]

27. Secondary Outcome: GMFR of SRH Antibody Response for Each Homologous Strain
Description: GMFR, the geometric mean of the ratio of GMTs (Day 21/Day 0), was measured using an SRH assay for homologous strains: H1N1 = A/Michigan/45/2015; H3N2 = A/Singapore/INFIMH-16-0019/2016; B/Colorado = B/Colorado/06/2017; B/Phuket = B/Phuket/3073/2013.
Time Frame: Baseline (Day 0), Day 21
Population: IPP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
Number analyzed (Participants) | 206 | 199
Ratio
  H1N1 | 1.7 [1.6 to 1.8] | 2.3 [2.1 to 2.5]
  H3N2 | 3.6 [2.9 to 4.4] | 2.5 [2.0 to 3.1]
  B/Colorado | 1.7 [1.5 to 1.9] | 2.0 [1.8 to 2.2]
  B/Phuket | 1.8 [1.6 to 2.1] | 2.4 [2.2 to 2.7]

ADVERSE EVENTS:
Time Frame: Day 0 (post-vaccination) up to ~9 months
Description: SAS. Participants that were non-compliant to protocol/GCP, as per investigator, were excluded from analysis.
Arm/Group | Quadrivalent (30 μg) VLP Vaccine | Active Comparator (Fluarix)
All-Cause Mortality (participants affected / at risk) | 12/6352 | 17/6366
Serious Adverse Events (participants affected / at risk) | 263/6352 | 266/6366
Other Adverse Events (participants affected / at risk) | 935/6352 | 908/6366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent (30 μg) VLP Vaccine (N=6352) | Active Comparator (Fluarix) (N=6366)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 4 (4)
Bursitis infective (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 2 (2)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 4 (4)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 20 (20) | 11 (12)
Pneumonia legionella (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Urosepsis (Infections and infestations) | 3 (3) | 0 (0)
Acral lentiginous melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Bronchial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Female reproductive neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoplasmacytoid lymphoma/immunocytoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic idiopathic pain syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 7 (7) | 9 (9)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
IVth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 5 (5)
Transient global amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 6 (6) | 3 (3)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0)
Corneal degeneration (Eye disorders) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 8 (8)
Angina pectoris (Cardiac disorders) | 3 (3) | 1 (1)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 11 (12) | 12 (13)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (5)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 5 (6) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 5 (5) | 3 (3)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 0 (0) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 2 (2)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypertensive crisis (Vascular disorders) | 3 (3) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 2 (2) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 3 (3)
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reactive gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Camptocormia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Lateral patellar compression syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (9) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hamartoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Syringomyelia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 4 (4)
Death (General disorders) | 1 (1) | 1 (1)
Incarcerated hernia (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Surgical failure (General disorders) | 1 (1) | 0 (0)
Vascular stent stenosis (General disorders) | 0 (0) | 1 (1)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal attack (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Fascial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Lacrimal structure injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Atrial appendage closure (Surgical and medical procedures) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quadrivalent (30 μg) VLP Vaccine (N=6352) | Active Comparator (Fluarix) (N=6366)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 12 (12) | 8 (8)
Cellulitis (Infections and infestations) | 1 (1) | 3 (3)
Conjunctivitis (Infections and infestations) | 2 (2) | 3 (3)
Cystitis (Infections and infestations) | 2 (2) | 6 (6)
Cystitis escherichia (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 2 (2)
Eye infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 8 (8)
Gastroenteritis viral (Infections and infestations) | 3 (3) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 2 (2)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0)
Genital infection fungal (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 1 (1)
Haemorrhagic fever with renal syndrome (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (1) | 3 (3)
Herpes zoster (Infections and infestations) | 5 (5) | 5 (5)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 13 (14)
Laryngitis (Infections and infestations) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Nasal herpes (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 88 (88) | 76 (77)
Onychomycosis (Infections and infestations) | 1 (1) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 5 (5) | 3 (3)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 2 (2) | 1 (1)
Pertussis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 4 (4) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4)
Respiratory tract infection (Infections and infestations) | 8 (8) | 5 (5)
Respiratory tract infection viral (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 9 (9) | 6 (6)
Root canal infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 13 (13) | 9 (9)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 52 (53) | 47 (48)
Urinary tract infection (Infections and infestations) | 15 (15) | 13 (13)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 3 (3)
Goitre (Endocrine disorders) | 0 (0) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 8 (8) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lipid metabolism disorder (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 8 (8)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 5 (5) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Fear (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2)
Listless (Psychiatric disorders) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (2)
Sleep disorder (Psychiatric disorders) | 2 (3) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 2 (2) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 3 (3)
Cerebral microangiopathy (Nervous system disorders) | 0 (0) | 1 (1)
Complex regional pain syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 19 (20) | 24 (25)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 61 (73) | 66 (71)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 2 (2) | 3 (3)
Movement disorder (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (3)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Posterior cortical atrophy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 2 (2) | 3 (3)
Sciatica (Nervous system disorders) | 2 (2) | 2 (2)
Sinus headache (Nervous system disorders) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 2 (2) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1) | 1 (3)
White matter lesion (Nervous system disorders) | 0 (0) | 1 (1)
Astigmatism (Eye disorders) | 0 (0) | 2 (2)
Binocular eye movement disorder (Eye disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1)
Blepharochalasis (Eye disorders) | 0 (0) | 1 (1)
Blindness transient (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Corneal warpage (Eye disorders) | 1 (1) | 0 (0)
Dry age-related macular degeneration (Eye disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Eye discharge (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 2 (2)
Eye swelling (Eye disorders) | 0 (0) | 2 (2)
Eyelid irritation (Eye disorders) | 0 (0) | 1 (1)
Eyelid margin crusting (Eye disorders) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1)
Eyelid pain (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 2 (2) | 1 (1)
Hyalosis asteroid (Eye disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 2 (2)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 1 (1) | 0 (0)
Neovascular age-related macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1)
Ocular rosacea (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 7 (7) | 7 (7)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 3 (3) | 4 (4)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 11 (11) | 11 (11)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3) | 0 (0)
Bundle branch block bilateral (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3) | 5 (5)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Dilatation atrial (Cardiac disorders) | 0 (0) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Left atrial dilatation (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 5 (5)
Mitral valve calcification (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 3 (3) | 4 (4)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2)
Pulmonary valve incompetence (Cardiac disorders) | 0 (0) | 2 (2)
Right atrial dilatation (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 5 (5)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 3 (3)
Aortic dilatation (Vascular disorders) | 0 (0) | 1 (1)
Aortic disorder (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 3 (4)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 35 (35) | 27 (27)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Microangiopathy (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 42 (42) | 46 (47)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 29 (31) | 30 (32)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 47 (47) | 41 (42)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 21 (22)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 17 (17)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 41 (42) | 56 (56)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 31 (33) | 25 (27)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 7 (7)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 8 (10)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 50 (53) | 53 (56)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 3 (3)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enlarged uvula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3) | 5 (5)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip erythema (Gastrointestinal disorders) | 0 (0) | 1 (2)
Lip pruritus (Gastrointestinal disorders) | 0 (0) | 1 (2)
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malocclusion (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 27 (27) | 30 (32)
Oesophageal food impaction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal motility disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Palatal oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 8 (8) | 6 (6)
Vomiting (Gastrointestinal disorders) | 13 (13) | 13 (14)
Biliary colic (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail bed disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10) | 8 (9)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 12 (12) | 8 (8)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (25) | 30 (30)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (21) | 26 (27)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (3)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 (11) | 12 (12)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 32 (34) | 35 (35)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 10 (10)
Nuchal rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 12 (12)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (14) | 11 (11)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 3 (3) | 4 (4)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 2 (2) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Renal cyst (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (4) | 7 (7)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 4 (4) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 3 (3) | 5 (5)
Chills (General disorders) | 15 (15) | 15 (15)
Discomfort (General disorders) | 2 (2) | 2 (2)
Face oedema (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 26 (27) | 32 (35)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Induration (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 8 (8) | 11 (11)
Injected limb mobility decreased (General disorders) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 4 (4)
Injection site erythema (General disorders) | 2 (2) | 3 (3)
Injection site haematoma (General disorders) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 12 (12) | 7 (7)
Injection site pruritus (General disorders) | 3 (3) | 4 (4)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 3 (3) | 5 (5)
Injection site warmth (General disorders) | 4 (4) | 2 (2)
Malaise (General disorders) | 11 (11) | 6 (6)
Mass (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 4 (4) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 9 (9) | 15 (16)
Swelling (General disorders) | 5 (5) | 6 (6)
Tenderness (General disorders) | 0 (0) | 1 (1)
Vaccination site haematoma (General disorders) | 1 (1) | 0 (0)
Vaccination site hypoaesthesia (General disorders) | 1 (1) | 0 (0)
Vaccination site induration (General disorders) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 1 (1)
Vaccination site pruritus (General disorders) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 3 (3)
Blood pressure increased (Investigations) | 13 (13) | 9 (9)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 2 (2)
Cardiac imaging procedure abnormal (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Thyroid hormones decreased (Investigations) | 0 (0) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 7 (7)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3) | 5 (6)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator understands that the information in the protocol is confidential and should not be disclosed, other than to those directly involved in the execution or the ethical review of the study, without prior written authorization from the Sponsor. It is, however, permissible to discuss information contained in the protocol with a participant in order to obtain consent once Institutional Review Board (IRB) approval is obtained.

DOCUMENTS (2):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT03739112/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/12/NCT03739112/SAP_001.pdf